CLINICAL TRIAL: NCT02995967
Title: Evaluation of Botulinum Toxin A Alone Versus Botulinum Toxin A With Hydrodistension for Treatment of Overactive Bladder
Acronym: HydrA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joseph Malek, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F160629005
Record Dates: First submitted 2016-12-09; First posted 2016-12-19 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin A alone group (Active Comparator): Just the intradetrusor injection of 100 units of botulinum toxin A alone
  Interventions: Drug: Botulinum toxin-A
- Hydrodistention group (Experimental): Hydrodistention at a pressure of 80 cm H2O for 5 minutes, prior to the intradetrusor injection of 100 units of botulinum toxin A
  Interventions: Procedure: Hydrodistention

INTERVENTIONS:
Procedure: Hydrodistention — The hydrodistention will then be performed with the bladder filled at a pressure of 80 cm H2O and noted to be full as evidenced by no further influx of water into the bladder. This volume will be held in the bladder for 5 minutes.
  Arms: Hydrodistention group
Drug: Botulinum toxin-A — Intradetrusor injection of 100 units of botulinum toxin a
  Arms: Botulinum toxin A alone group

SUMMARY:
The specific aim of this trial is to determine if hydrodistention at the time of intradetrusor injection of botulinum toxin A has additional benefit in patients with refractory overactive bladder (OAB) and urgency symptoms compared to intradetrusor injection of botulinum toxin A alone.

Consented patients will be randomized to hydrodistention at a pressure of 80 cm H2O for 5 minutes, prior to the intradetrusor injection of 100 units of botulinum toxin A (hydrodistention group) or intradetrusor injection of 100 units of botulinum toxin A alone (botulinum toxin A alone group).

The primary aim will be subjective improvement measured as change from baseline at 12 weeks using the OAB-q bother subscale.

ELIGIBILITY:
Inclusion Criteria:

* Women with refractory overactive bladder symptoms, failing a credible behavioral therapy intervention and medical therapy or not tolerating medical therapy. Patients who are on medical therapy will stop the medical therapy for at least 2 weeks prior to botulinum toxin A treatment in the study
* Female ≥ 18 years old
* Desires further treatment for OAB symptoms.
* Express understanding and ability to perform clean intermittent self-catheterization (CISC) if required.
* Ability to consent
* Ability to complete all study related items and interviews

Exclusion Criteria:

* Post void residual urine volume > 150 mL as assessed by catheter or ultrasound
* History of intradetrusor botulinum toxin A injection
* History of or current cancer of the genitourinary or gynecology tract
* Neurogenic bladder
* Interstitial cystitis
* Current urinary tract infection (can be treated and re-considered for study)
* Current active sacral neuromodulation device
* Non-English speaking
* History of chronic pelvic pain
* Hematuria not previously evaluated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama Birmingham Hospital, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 3 participants completed the study, no analysis done due to study being stopped for poor enrollment.
Groups:
- Botulinum Toxin A Alone Group: Intradetrusor injection of 100 units of botulinum toxin A alone
  Botulinum toxin-A: Intradetrusor injection of 100 units of botulinum toxin a
Period: Overall Study
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Customized [Count of Participants; unit: Participants]
  age over 50 yrs | 1 | 2 | 3
  age uner 50 yrs | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or AlaskaNative | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Symptom Bother
Description: The primary outcome will be measured as change from baseline at 12 weeks using the OAB-q bother subscale which consists of eight questions assessing symptom bother with a possible score from 0 to 100 with a higher score indicating greater symptom bother.
Time Frame: 12 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Urge Urinary Incontinence Episodes
Description: Number of UUI episodes as reported in a 3-day bladder diary at 12 weeks as measured in change from baseline.
Time Frame: 12 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Total Number of Voids
Description: Total number of voids reported in the 3-day bladder diary at 12 weeks as measured in change from baseline.
Time Frame: 12 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Subjects Requiring Clean Intermittent Self-catheterization
Description: Proportion of subjects requiring clean intermittent self-catheterization (CISC) post-operatively as reported at 2 week post-operative visit. CISC will be initiated at post-void residual volumes of > 300 mL or > 150 mL in the presence of bothersome retention symptoms.
Time Frame: 2 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Post Void Residual Volume
Description: Post-void residual volume (PVR) at the 2 week follow-up visit measured with catheter or bladder scan.
Time Frame: 2 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Rate of UTI
Description: Rate of urinary tract infection (UTI) as assessed by positive urine culture in patients having symptoms (dysuria, urgency, frequency, temperature ≥ 38 degrees Celcius, and/or suprapubic pain) at the 2 weeks post-operative visit. Subjects who call throughout the study complaining of symptoms but are unable to give a urine culture in clinic will also be treated and reported as having had a UTI.
Time Frame: 2 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Quality of Life Measures
Description: Health related quality of life (HRQL) will be measured as a change from baseline at 12 weeks using the OAB-q HRQL subscale part which consists of 25 questions that assess HRQL addressing coping, concern, sleep, and social interaction where the scoring scale is from 0 to 100 with a higher score indicating a better quality of life.
Time Frame: 12 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient Impression of Improvement
Description: Patient global impression of improvement at 12 weeks as measured using the Patient Global Impression of Improvement Questionnaire (PGI-I).
Time Frame: 12 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction at 12 weeks as measured using Patient Satisfaction Questionnaire (PSQ).
Time Frame: 12 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Quality of Life Measures
Description: Subjective outcome at 24 weeks using the OAB-q
Time Frame: 24 weeks
Population: No analysis done due to study being stopped for poor enrollment
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Botulinum Toxin A Alone Group | Hydrodistention Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02995967/Prot_SAP_000.pdf